CLINICAL TRIAL: NCT04689958
Title: The Benefits of Vitamin D 5000 IU as Add on Therapy in the Management of Painful Diabetic Neuropathy Patient: Randomized Clinical Trial
Brief Title: The Benefits of Vitamin D 5000 IU as Add on Therapy in the Management of Painful Diabetic Neuropathy Patient
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Duta Wacana Christian University (Other)
Collaborators: PT SOHO Global Health Tbk (Unknown)
Responsible Party: Principal Investigator, Rizaldy Taslim Pinzon, Principal investigator, Neurologist, Duta Wacana Christian University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VITAMIND5000IU
Record Dates: First submitted 2020-12-19; First posted 2020-12-30 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Painful Diabetic Neuropathy
Keywords: Vitamin D; Standard therapy; Neuropathy; Diabetic neuropathy
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Standard of Care; Vitamin D; Tablets

STUDY DESIGN:
Intervention Model Description: Eligible subjects were randomly allocated to receive any of the following regiments: standard therapy consists of pregabalin, gabapentine, or amitriptyline (control group) or standard therapy and vitamin D 5000 IU tablet once daily (experimental group).
Masking Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Receive standard therapy consists of gabapentin, pregabalin, or amitriptyline and vitamin D 5000 IU once daily (experimental group).
  Interventions: Drug: Standard therapy; Drug: Vitamin D 5,000IU Oral Tablet
- Control Group (Active Comparator): Receive standard therapy consists of gabapentin, pregabalin, or amitriptyline
  Interventions: Drug: Standard therapy

INTERVENTIONS:
Drug: Standard therapy — Gabapentin, pregabalin, or amitriptyline
Drug: Vitamin D 5,000IU Oral Tablet — Vitamin D 5000 IU oral tablet once daily
  Arms: Experimental Group

SUMMARY:
Diabetic neuropathy is one of the micro-vascular complications of diabetes, 30-50% occurring in all diabetic patients. This complication is one of the major cause of morbidity and mortality in diabetic patientsand leading to a deterioration of their quality life. A deficiency of vitamin D [25-hydroxyvitamin D, 25(OH) D] is common in patient with diabetes and low concentrations are associated with the presence and severity of sensory neuropathy in diabetes. Vitamin D deficiency has been shown to be an independent risk factor for diabetic peripheral neuropathy (DPN). Topical and oral vitamin D have been reported significantly reduce the symptoms and the pain of DPN. However, no case control clinical trial have been reported that demonstrate the efficacy of vitamin D supplementation on the symptoms of DPN.

Painful in diabetic neuropathy is a major complication of diabetes, characterized by pain, tingling, burning and cramps in the lower legs and feet with a signification reduction in quality of life. Recently, there shown a significant reduction in the severity of painful diabetic neuropathy after treatment with vitamin D. Patient with diabetes have a poor quality of life compared to person without diabetes. The current study assessed the benefits of add on oral vitamin D 5000 IU on diabetic neuropathy patient to pain impact in daily life.

DETAILED DESCRIPTION:
This was randomized clinical trial, active comparator, open label, controlled study from the period of November 2020 - November 2021 at Bethesda Hospital, Yogyakarta, Indonesia.

There were 60 painful diabetic neuropathy patients who fulfilled the inclusion and exclusion criteria. Each subject had been followed up from the first day of medication administration until 8 weeks after medication administration.

Ethical approval number ((kosong)) was obtained from Health Research Ethics Committee, Bethesda Hospital Yogyakarta.

The hypothesis of this study:

a. Add on oral vitamin D 5000 IU to standard treatment in patients with painful diabetic neuropathy is more effective in reducing pain and neuropathic symptoms in 8 weeks of treatment compared with standard treatment, b. Add on oral vitamin D 5000 IU to standard treatment in patients with painful diabetic neuropathy is as safe as standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Adult age (>18 years old)
* Diagnosed as painful diabetic neuropathy based on validated Diabetic Neuropathy Symptoms (DNS) and Diabetic Neuropathy Examination (DNE)
* Low vitamin D status of <30 ng/ml

Exclusion Criteria:

* Subjects with significant renal and liver problem
* Subjects with known hypersensitivity to vitamin D 5000 IU
* Pregnancy and breastfeeding patients
* Patients that enrolled any clinical trial within a month
* Not competent enough in giving approval and answering questionnaires

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-11-03 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Improvement in Visual Analogue Scale (VAS) at week 4 | 4 weeks after treatment initiation
  Change in pain impact on daily life as measured by Visual Analogue Scale (VAS) from its baseline value. Visual analogue scale is a continuous scale comprised of a horizontal or vertical line, usually 10 centimeters (100 mm) in length, anchored by 2 verbal descriptors, one for each symptom extreme. The scale is most commonly anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100). The respondent is asked to place a line perpendicular to the VAS line at the point that represents their pain intensity. Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.
Improvement in Visual Analogue Scale (VAS) at week 8 | 8 weeks after treatment initiation
  Change in pain impact on daily life as measured by Visual Analogue Scale (VAS) from its baseline and week 4 value. Visual analogue scale is a continuous scale comprised of a horizontal or vertical line, usually 10 centimeters (100 mm) in length, anchored by 2 verbal descriptors, one for each symptom extreme. The scale is most commonly anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100). The respondent is asked to place a line perpendicular to the VAS line at the point that represents their pain intensity. Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.
Improvement in Numeric Pain Scale at week 4 | 4 weeks after treatment initiation
  Change in pain impact on daily life as measured by Numeric Pain Scale from its baseline value. Numeric pain scale is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. Higher scores indicating greater pain intensity.
Improvement in Numeric Pain Scale at week 8 | 8 weeks after treatment initiation
  Change in pain impact on daily life as measured by Numeric Pain Scale from its baseline and week 4 value. Numeric pain scale is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. Higher scores indicating greater pain intensity.
Improvement in Brief Pain inventory at week 4 | 4 weeks after treatment initiation
  Change in pain impact on daily life as measured by Brief Pain Inventory from its baseline value. The Brief Pain Inventory evaluates a patient's pain experience through a number of different scales. There are line drawings of the front and back of a human body on which patients mark the location of their pain. Patients are asked to list the treatments or medications that they are using and how much relief they have provided in the past 24 hours. In addition, patients fill out 11 different numeric rating scale that ask about pain intensity (ranging from 0 to 10) and the effect of the pain on their ability to function during various activities of daily living. A higher score indicates greater pain intensity.
Improvement in Brief Pain inventory at week 8 | 8 weeks after treatment initiation
  Change in pain impact on daily life as measured by Brief Pain Inventory from its baseline and week 4 value. The Brief Pain Inventory evaluates a patient's pain experience through a number of different scales. There are line drawings of the front and back of a human body on which patients mark the location of their pain. Patients are asked to list the treatments or medications that they are using and how much relief they have provided in the past 24 hours. In addition, patients fill out 11 different numeric rating scale that ask about pain intensity (ranging from 0 to 10) and the effect of the pain on their ability to function during various activities of daily living. A higher score indicates greater pain intensity.

CONTACTS AND LOCATIONS:
Overall Officials: Rizaldy T Pinzon, MD, MSc, PhD, Principal Investigator — Duta Wacana Christian University
Locations (1):
- Bethesda Hospital Yogyakarta, Yogyakarta, Special Region of Yogyakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ghadiri-Anari A, Mozafari Z, Gholami S, Khodaei SA, Aboutorabi-Zarchi M, Sepehri F, Nadjarzade A, Rahmanian M, Namiranian N. Dose vitamin D supplementations improve peripheral diabetic neuropathy? A before-after clinical trial. Diabetes Metab Syndr. 2019 Jan-Feb;13(1):890-893. doi: 10.1016/j.dsx.2018.12.014. Epub 2018 Dec 20. PMID 30641826
- [Background] Shehab D, Al-Jarallah K, Abdella N, Mojiminiyi OA, Al Mohamedy H. Prospective evaluation of the effect of short-term oral vitamin d supplementation on peripheral neuropathy in type 2 diabetes mellitus. Med Princ Pract. 2015;24(3):250-6. doi: 10.1159/000375304. Epub 2015 Feb 26. PMID 25720672
- [Background] Shehab D, Al-Jarallah K, Mojiminiyi OA, Al Mohamedy H, Abdella NA. Does Vitamin D deficiency play a role in peripheral neuropathy in Type 2 diabetes? Diabet Med. 2012 Jan;29(1):43-9. doi: 10.1111/j.1464-5491.2011.03510.x. PMID 22050401
- [Background] Soderstrom LH, Johnson SP, Diaz VA, Mainous AG 3rd. Association between vitamin D and diabetic neuropathy in a nationally representative sample: results from 2001-2004 NHANES. Diabet Med. 2012 Jan;29(1):50-5. doi: 10.1111/j.1464-5491.2011.03379.x. PMID 21726279
- [Background] Valensi P, Le Devehat C, Richard JL, Farez C, Khodabandehlou T, Rosenbloom RA, LeFante C. A multicenter, double-blind, safety study of QR-333 for the treatment of symptomatic diabetic peripheral neuropathy. A preliminary report. J Diabetes Complications. 2005 Sep-Oct;19(5):247-53. doi: 10.1016/j.jdiacomp.2005.05.011. PMID 16112498
- [Background] Lee P, Chen R. Vitamin D as an analgesic for patients with type 2 diabetes and neuropathic pain. Arch Intern Med. 2008 Apr 14;168(7):771-2. doi: 10.1001/archinte.168.7.771. No abstract available. PMID 18413561
- [Background] Bell DS. Reversal of the Symptoms of Diabetic Neuropathy through Correction of Vitamin D Deficiency in a Type 1 Diabetic Patient. Case Rep Endocrinol. 2012;2012:165056. doi: 10.1155/2012/165056. Epub 2012 Dec 12. PMID 23304571
- [Background] Basit A, Basit KA, Fawwad A, Shaheen F, Fatima N, Petropoulos IN, Alam U, Malik RA. Vitamin D for the treatment of painful diabetic neuropathy. BMJ Open Diabetes Res Care. 2016 Feb 10;4(1):e000148. doi: 10.1136/bmjdrc-2015-000148. eCollection 2016. PMID 27026808
- [Background] Alam U, Fawwad A, Shaheen F, Tahir B, Basit A, Malik RA. Improvement in Neuropathy Specific Quality of Life in Patients with Diabetes after Vitamin D Supplementation. J Diabetes Res. 2017;2017:7928083. doi: 10.1155/2017/7928083. Epub 2017 Dec 28. PMID 29445752
- [Derived] Pinzon RT, Wijaya VO, Veronica V. The Benefits of Add-on Therapy of Vitamin D 5000 IU to the Vitamin D Levels and Symptoms in Diabetic Neuropathy Patients: A Randomized Clinical Trial. J Pain Res. 2021 Dec 19;14:3865-3875. doi: 10.2147/JPR.S341862. eCollection 2021. PMID 34984028